CLINICAL TRIAL: NCT06336564
Title: Microablative Radiofrequency in the Treatment of Urinary Symptoms Associated With Genitourinary Syndrome of Menopause: Randomized Clinical Trial
Brief Title: Microablative Radiofrequency in the Treatment of Urinary Symptoms Associated With Genitourinary Syndrome of Menopause
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Principal Investigator, Patricia Lordelo, Head of the CentroAAP, Centro de Atenção ao Assoalho Pélvico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 71168623.6.0000.5544
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Menopause; Urinary Incontinence
Keywords: Genitourinary syndrome of menopause; Microablative Radiofrequency
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Pelvic floor muscle training
  Interventions: Other: Pelvic floor muscle training
- Intervention Group (Experimental): Pelvic floor muscle training and microablative radiofrequency
  Interventions: Other: Pelvic floor muscle training; Device: Microablative Radiofrequency

INTERVENTIONS:
Other: Pelvic floor muscle training — Verbal information will be given about location, function and the correct way to contract the pelvic floor muscles (PFM). Participants will be instructed on how to perform "The Knack", which is a pre-contraction of the PFM during some abdominal effort, such as coughing, sneezing or laughing. The exercises consist of two series of 10 maximum contractions sustained for 5 seconds and 10 seconds of relaxation and two series of 10 maximum rapid contractions with two seconds of maintenance and four seconds of relaxation, with one minute of rest between each series. Participants will be instructed to perform the same exercises at home (twice a day) and to fill out a training diary, allowing researchers to monitor and check whether the exercises are actually being performed. The protocol will be repeated with the researcher three times in total, every 30 to 40 days.
Device: Microablative Radiofrequency — Patients will be placed in the lithotomy position and through speculum examination and under direct vision or guided by colposcope, sequential application of radiofrequency will be carried out on the vaginal walls and introitus. The Wavetronic 6000 Touch device will be used with the Megapulse HF FRAXX system (Loktal Medical Electronics, São Paulo, Brazil), equipped with an electronic energy fractionation circuit, connected to a vaginal pen with 64 microneedles, 200μm in diameter and 1 mm in length, mounted on a Teflon body and divided into a matrix of eight columns with eight needles each. In the vestibule and vaginal opening, 10% lidocaine spray will be applied three minutes before the procedure. Three applications will be carried out in the vagina/vaginal introitus, with an interval of 30 to 40 days.
  Arms: Intervention Group

SUMMARY:
Genitourinary Syndrome fo Menopause (GSM) is made up of a set of changes in the region of the vulva, vagina and lower urinary tract associated with a decrease in estrogen levels in the urogenital tissue, which leads to a reduction in blood supply, disorders in collagen metabolism and skin elasticity. The standard treatment for urinary incontinence during menopause is pelvic floor muscle training, associated or not with local hormone replacement therapy. Although low cost and easy to access, it is associated with low patient's adherence. Physical methods such as laser and radiofrequency in non-ablative, ablative and microablative forms are technologies that have recently been used in the vaginal mucosa to promote neoelastogenesis and neocollagenesis. It is hypothesized that menopausal women, who present symptoms of GSM, may benefit from this new, minimally invasive resource (microablative radiofrequency). This is a randomized clinical trial in which women aged between 40 and 65 years old will be included with clinical complaints of urinary symptoms associated with GSM. A basic anamnestic questionnaire will be used as the study instrument to collect sociodemographic, clinical data and symptoms, following the routine and standard of the service. To evaluate the treatment, the following will be used: voiding diary, pad test, vaginal cytology, histopathology, Female Sexual Function Index (FSFI), Short-Form Health Survey - SF-36 Questionnaire, King's Health Questionnaire, evolution of symptoms (dryness, pain during sexual activity, vaginal laxity, itching, burning sensation and pain in the vaginal introitus) and level of patient's satisfaction. Patients will be randomized into: group 1 or control group, which will perform pelvic floor muscle training, PFMT, with supervision (three times) and at home twice a day, and group 2 or test group, which will perform the same PFMT protocol associated with vaginal microablative radiofrequency. 10% lidocaine spray will be applied three minutes before the procedure and three applications will be made to the vagina/vaginal introitus, with an interval of 30 to 40 days. The purpose of this study is to test the efficacy and duration of effect of microablative radiofrequency in the treatment of urinary symptoms associated with GSM.

ELIGIBILITY:
Inclusion Criteria:

* Clinical complaint of urinary incontinence associated to Genitourinary Syndrome of Menopause.
* Negative cervical oncotic cytology, within the last 3 years.

Exclusion Criteria:

* Patients with cognitive deficit;
* Patients with chronic degenerative neurological diseases;
* Post-void residue greater than 50 ml;
* Carriers of a pacemaker and implantable cardioverter defibrillator;
* Use of hormonal therapy (topical or systemic) starting in the 2 months prior to the initial assessment;
* Patients undergoing brachytherapy or pelvic radiotherapy;
* Patients that had reconstructive pelvic surgery;
* Pregnant women.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Resolution or improvement of episodes of urinary loss assessed by pad test | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment.
  Participants will perform the one-hour Pad Test to diagnose and quantify urinary loss. Initially, the absorbent will be placed in a closed plastic bag and weighed on a precision electronic scale (Denver Instrument®). Then, the participant will be instructed to put on the pad, drink 500 ml of water in a maximum of 15 minutes and remain at rest for another 15 minutes, this phase represents 30 minutes of the test. In the other 30 minutes, the participant will be asked to perform certain standardized activities simulating activities of daily life (going up and down stairs, sitting down and standing up ten times, coughing ten times, picking up objects from the floor five times, running in the same place for one minute and washing the hands under running water for one minute).
Resolution or improvement of episodes of urinary loss assessed by urinary diary | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment
  Participants will be instructed to keep a voiding diary at home for three days to record water intake, urinary volume and the number of incontinence episodes, as well as episodes of urgency and nocturnal enuresis.
Number of patients with tolerability related to treatment assessed by Likert Scale. | At each of the three sessions (every 30 to 40 days), 30 days after the end of treatment and 12 months after the end of the treatment.
  Likert scale of 3 points will be asked to the patients: 1) impossible to tolerate the treatment, 2) not nice, but possible to tolerate, 3) very tolerable.
Number of patients with adverse effects related to treatment assessed by histopathology. | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment.
  To evaluate the safety in tissue effect of FRAXX, samples of vaginal tissue will be obtained through a biopsy taken from the lateral walls, in the middle third of the vagina, for histopathological study. Procedure carried out under colposcopic vision, using a 3mm loop attached to the radiofrequency device, "surgery" mode, removing a small vaginal fragment.
Resolution or improvement of episodes of urinary loss assessed by questionnaire. | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment.
  The questionnaire to be used will be International Consultation on Incontinence Questionnaire- Short Form (ICIQ-SF) which is a self-administered questionnaire that assesses the impact of UI on quality of life and the classification of urinary loss. The ICIQ-SF is composed of four questions that assess the frequency, severity and impact of UI, in addition to a set of eight self-diagnosis items, related to the causes or situations of UI experienced by patients. The higher the score, the greater the severity of urinary incontinence and the greater the impact on the patient's quality of life.

SECONDARY OUTCOMES:
Recovery of vaginal health assessed by Vaginal Index Maturation | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment
  The cytological evaluation will be carried out using a vaginal smear collected from the lateral vaginal wall with a spatula ; the percentage of superficial (%S), intermediate (%I) and parabasal (P%) cells are counted and the mucosa is then classified according to the Vaginal Maturation Index (VMI) of the Meisel formula [(1, 0 x %S) + (0.5 x %I) + (0.0 x %P)] as atrophic, hypotrophic or eutrophic.
Recovery of vaginal health assessed by vaginal pH | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment
  Vaginal pH will be measured with a pH indicator strip between 0 and 14 (MColorpHastTM, Merck, Germany), placed in contact with the mucosa of the middle third of the vaginal canal, with the help of a speculum.
Improvement of Sexual Function assessed by Female Sexual Function Index | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment
  A self-administered questionnaire, which proposes to evaluate female sexual response in the domains: sexual desire, sexual arousal, vaginal lubrication, orgasm, sexual satisfaction and pain. It presents 19 questions that assess sexual function in the last four weeks and presents scores for each component. For each question there is a response pattern, between 0 and 5 in an increasing order, except for questions about pain, where the score is reversed. The domain that presents a score equal to zero means that the interviewee did not report sexual intercourse in the last four weeks. Individual scores are obtained by summing the items that comprise each domain (simple score), which are multiplied by the factor of that domain and provide the weighted score. The final score (total score: minimum of 2 and maximum of 36) is obtained by adding the weighted scores for each domain. The cut-off is: > or = 26 points - no sexual dysfunction; bellow 26 - sexual dysfunction.
Improvement of quality of life assessed by Short-Form Health Survey (SF-36) | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment
  It consists of 36 items that encompass 8 domains: functional capacity, physical aspects, pain, general health, vitality, social aspects, emotional aspects and mental health. It presents a final score from 0 to 100, where zero represents the worst general health status and 100 the best general health status.
Improvement or resolution of urinary incontinence and the impact on quality of life assessed by King's Health Questionnaire. | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment
  It consists of 21 questions and has four to five answer options on the LIKERT scale. It involves nine domains: general health perceptions, impact of incontinence, function restrictions, physical limitations, social limitations, personal relationships, emotions, sleep and energy, and severity measures. Furthermore, it has an independent scale called Symptom Severity Scale, which contains 11 items, measuring the presence and severity of urinary symptoms. The score, both per domain and its global score, is obtained from a minimum of 0 (best quality of life) to a maximum of 100 (worst quality of life).
Degree of patient satisfaction using a five-point Likert scale. | Before the beginning of the treatment, 30 days after the end of treatment and 12 months after the end of the treatment
  It will classify patient's level of satisfaction as: 1) very dissatisfied; 2) dissatisfied; 3) unchanged; 4) satisfied; 5) very satisfied.
Evolution of vaginal symptoms assessed by Visual Analogue Scale (VAS) | Immediately after the initial physical examination and at the end of each of the three session (every 30 to 40 days).
  Intensity of vaginal symptoms (dryness, pain during sexual activity, vaginal laxity, itching, burning sensation and pain in the vaginal introitus) will be asked to the participants. VAS is divided from 0 to 10 points. 0 will be considered as absence of the symptom and 10 will represent the maximum possible symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Lordelo, PhD, Principal Investigator — Pelvic Floor Care Center
Locations (1):
- Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No